CLINICAL TRIAL: NCT04003480
Title: Prospective, Multicenter Study Evaluating the Performance and Safety of FRAME, External Support for Lower Limb Autologous Grafts.
Brief Title: FRAME, External Support for Lower Limb Autologous Grafts
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: no patients have been enrolled. Study suspended due to change of sponsor priorities during COVID
Sponsor: Vascular Graft Solutions Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CD0177
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Peripheral Arterial Disease; Peripheral Artery Disease
Keywords: Saphenous vein graft; PAD; Peripheral bypass surgery; external support
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- FRAME (Experimental): Vein graft to be treated with FRAME
  Interventions: Device: FRAME

INTERVENTIONS:
Device: FRAME — External support for vein grafts in peripheral bypass surgery

SUMMARY:
30 patients will be enrolled in a prospective, multi-center, one-arm study, enrolling patients with claudication and chronic limb ischemia scheduled for lower limb venous bypass grafting on clinical grounds with single segment autologous saphenous vein.

Subjects will be followed for 5 years, with follow up visits at 1, 3, 6, 12 months, 2, 3, 4, 5, years post operation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient scheduled for infrainguinal peripheral artery bypass surgery with single segment autogenous saphenous vein.
2. Rutherford classification 3-6
3. Adequate revascularization target defined as an infrainguinal arterial segment distal to the area of stenosis/occlusion which can support a distal anastomosis of a surgical bypass.
4. Patient is able and willing to give their informed written consent.
5. Patient is able and willing to comply with study follow up requirements.
6. Patient is ≥ 18 years of age

Exclusion Criteria:

1. Patients indicated for endovascular treatment
2. Prior surgical bypass procedure in ipsilateral lower limb.
3. Active ulcer/infection/gangrene at the intended distal anastomosis site.
4. Severe vein varicosity
5. Saphenous vein with external pressurized diameter of less than 3.5 mm or more than 8 mm.
6. Spliced vein technique
7. In-situ vein technique
8. Pedal/plantar distal anastomosis
9. Planned above ankle amputation on ipsilateral limb within 4 weeks of index procedure.
10. Patients with history of hypercoagulable conditions.
11. Patients with significant stenoses distal to the planned anastomotic site and any other known conditions that could adversely affect graft patency.
12. Concomitant life-threatening disease likely to limit life expectancy to less than 2 years.
13. Contraindication to recommended study medications
14. Participating in any other investigational study for either drug or device which can influence collection of valid data under this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-12-31 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 12 months
  Freedom of vein graft from occlusion and clinically driven target lesion revascularization as measured by Doppler Ultrasound

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Lutheran Hospital of Indiana, Fort Wayne, Indiana
  - University of Maryland Baltimore, Baltimore, Maryland
  - Mount Sinai Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No